CLINICAL TRIAL: NCT00385502
Title: A Phase II Trial of the Safety, Local Tolerability, and Efficacy of EcoNail™ (Econazole 5%/SEPA® 18% Nail Lacquer) in Onychomycosis of the Great Toenail
Brief Title: A Trial of the Safety and Efficacy of EcoNail™ in the Treatment of Fungus Infections of the Great Toenail
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abeona Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCHM EC-200
Record Dates: First submitted 2006-10-05; First posted 2006-10-09 (Estimated); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Onychomycosis
Keywords: toenail; fungus; onychomycosis; antifungal; anti-fungal; nail
MeSH Terms: conditions — Onychomycosis | interventions — Econazole; Separase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EcoNail™ (Experimental): econazole 5%/SEPA® 18% nail lacquer
  Interventions: Drug: EcoNail™ (econazole 5%/SEPA® 18% nail lacquer)

INTERVENTIONS:
Drug: EcoNail™ (econazole 5%/SEPA® 18% nail lacquer) — nail lacquer applied daily for 48 weeks
  Other Names: econazole; SEPA

SUMMARY:
Approximately 40 qualified subjects with mild-to-moderate great toenail fungus infection will be treated for 48 weeks with lacquer application to at least one affected great toenail. All subjects will receive treatment with EcoNail™ lacquer.

DETAILED DESCRIPTION:
This study will use a multi-center, open-label study design in subjects with onychomycosis of at least one great toenail to assess the safety, local tolerability, and efficacy of chronic daily ungual application of EcoNail™. Forty (40) evaluable subjects will apply study drug daily to at least one affected great toenail for 48 weeks. The subjects must comply with all inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are men and women greater than or equal to 18 years of age and less than or equal to 65 years of age.
* Female subjects who are post-menopausal (amenorrheic for at least 1 year), surgically sterile, have a partner with a vasectomy, or routinely using an acceptable means of contraception (acceptable methods may include hormonal contraceptives, intrauterine device, spermicide and barrier, abstinence and partner/spouse sterility).
* Subjects who have mycologically confirmed distal subungual onychomycosis of at least one or both great toenails ("target toenails"), defined as a positive result by office-based KOH preparation (± Chlorazol B) and by laboratory culture demonstrating one of more of the following organisms: T. rubrum, T. mentagrophytes, T. tonsurans and/or E. floccosum
* Subjects who have target toenail showing 20-65% (+/- 2%) involvement as judged by the clinical investigator.
* Subjects who have target toenail showing great than or equal to 3 mm distal involvement as judged by the clinical investigator.
* Subjects who have target toenail showing great than or equal to 2 mm proximal clear nail at the cuticle.
* Subjects must agree not to apply other nail polish or related products to the affected nails for the duration of the study.
* Subjects must refrain from filing, clipping, or otherwise disturbing the treated nail(s) for the duration of the study [NOTE: Clinic personnel will debride the affected nails during monthly visits. Subjects should not engage in these activities at home during the course of the study.]
* Subjects must have the ability to understand the nature of the study and any hazards of participating in it and the willingness to communicate satisfactorily with the investigator and staff and to participate in, and comply with the requirements of the entire study.
* Subjects must be able to read and sign the study Informed Consent form and comply with the requirements outlined in the informed consent form.

Exclusion Criteria:

* Subjects with < 20% or > 65% (+/- 2%) involvement of the target toenail.
* Subjects with great than or equal to 4 mm thickness of the target toenail.
* Subjects with totally dystrophic great toe.
* Subjects with great toenails which show white superficial or proximal subungual onychomycosis, or a "spike" of onychomycosis extending to the cuticle.
* Subjects whose nail cultures grow Candida species as the only pathogen.
* Subjects who have reported treatment with a topical anti-fungal agent for onychomycosis during the four weeks prior to screening for this study.
* Subjects who have been treated with a systemic anti-fungal agent during the three months prior to screening for this study.
* Subjects with any other nail abnormality or dermatological condition, including (but not limited to) psoriasis and lichen planus, that could prevent obtaining a normal-appearing toenail if complete cure was achieved or could otherwise interfere with required study assessments.
* Subjects with a history of organ transplantation, Human Immunodeficiency Virus (HIV) seropositivity or other historical or clinical evidence of an immunocompromised state.
* Subjects with a history of uncontrolled insulin-dependent diabetes mellitus.
* Subjects with a history of diabetic peripheral neuropathy.
* Subjects with a history of clinically significant lower extremity peripheral occlusive vascular disease.
* Subjects with a presence of plantar (moccasin) tinea pedis.
* Subjects with a history of hypersensitivity or allergic reactions on the skin or nails, including reactions to nail polish and/or nail polish remover.
* Subjects known to have an allergy to econazole, ethanol, Eudragit, or SEPA.
* Female subjects who are pregnant or lactating.
* Subjects with clinically relevant abnormal history, physical findings, or laboratory values at the screening assessment that could interfere with the objectives or the safety of the volunteer.
* Subjects who have a condition or abnormality that in the investigator's opinion may interfere with the assessments, conduct of the study, may affect the subject's safety, or is otherwise unsuitable for enrollment.
* Subjects who are currently participating or, within the previous 30 days, have participated in another investigational drug study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-09 (Actual); Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Determine effectiveness of EcoNail™ lacquer, as determined by effects on nail mycology and appearance, when applied daily for 48 weeks to diseased great toenails in subjects with onychomycosis. | Week 48

SECONDARY OUTCOMES:
Evaluate the safety and local tolerability of EcoNail™ lacquer under the same circumstances. | Week 56

CONTACTS AND LOCATIONS:
Overall Officials: Michael H. Silverman, MD, Study Director — Biostrategics Consulting, Ltd.
Locations (3):
- United States (3):
  - Tucson, Arizona
  - New York, New York
  - Portland, Oregon

REFERENCES:
- See also: Sponsor's website — http://www.accesspharma.com/index.shtml